CLINICAL TRIAL: NCT01103648
Title: Synergistic Effect of Simvastatin and Ezetimibe on Lipid and Pro-inflammatory Profiles in Pre-diabetic Subjects
Brief Title: Effect of Simvastatin and Ezetimibe on Lipid and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Sandra Roberta Gouvea Ferreira, Federal University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUSaoPaulo
Record Dates: First submitted 2010-04-12; First posted 2010-04-15 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2007-11

CONDITIONS: Prediabetes; Hypercholesterolemia; Inflammation; Cardiovascular Risk
Keywords: Prediabetes; Statin; Ezetimibe; Pleiotropic effects; Cardiometabolic risk
MeSH Terms: conditions — Prediabetic State; Hypercholesterolemia; Inflammation | interventions — Simvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe; Hypolipidemic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Simvastatin arm (Active Comparator): A subset of individuals started the study period taking monotherapy with simvastatin. After a 12-week period, ezetimibe was combined to the initial monotherapy for more 12 weeks (combination period = experimental).
  Interventions: Drug: Simvastatin
- Ezetimibe arm (Active Comparator): A subset of individuals started the study period taking monotherapy with ezetimibe. After a 12-week period, simvastin was combined to the initial monotherapy for more 12 weeks (combination period = experimental).
  Interventions: Drug: Ezetimibe
- Simvastatin-Ezetimibe arm (Experimental): To each subset of individuals which started the study period taking monotherapy with simvastatin or ezetimibe (active comparators), the other drug (ezetimibe or simvastatin, respectively) was combined for more 12 weeks (combination period = experimental arm).
  Interventions: Drug: Combination Simvastatin plus Ezetimibe

INTERVENTIONS:
Drug: Simvastatin — Tablets of simvastatin 20 mg administered once a day for 12 weeks
  Other Names: Statin
  Arms: Simvastatin arm
Drug: Ezetimibe — Tablets of ezetimibe 10 mg administered once a day for 12 weeks
  Other Names: Lipid-lowering drug
  Arms: Ezetimibe arm
Drug: Combination Simvastatin plus Ezetimibe — Simvastatin 20 mg, once a day, was administered for an additional 12-week period for the subset of individuals who took the initial monotherapy with ezetimibe 10 mg (12 week duration).
  Ezetimibe 10 mg, once a day, was administered for an additional 12-week period for the subset of individuals who took the initial monotherapy with simvastatin 20 mg (12 week duration).
  This Combination represents the experimental period of the present study.
  Other Names: Simvastatin; Statin; Ezetimibe; Lipid-lowering drugs
  Arms: Simvastatin-Ezetimibe arm

SUMMARY:
Ezetimibe specifically blocks the absorption of dietary and biliary cholesterol and plant sterols. Synergism of ezetimibe-statin therapy on LDL-cholesterol has been demonstrated, but data concerning the pleiotropic effects of this combination are controversial. We tested the hypothesis that the combination of simvastatin and ezetimibe would induce improvement in inflammatory status, as reflected by leukocyte count and CRP, IL-6 and TNF-a levels. This open-label trial evaluated whether this combination results in a synergistic effect the pro-inflammatory status of pre-diabetic subjects. Fifty pre-diabetic subjects were randomly assigned to one of 2 groups, one receiving ezetimibe (10 mg/d), the other, simvastatin (20 mg/d) for 12 weeks, followed by an additional 12-week period of combined therapy.

DETAILED DESCRIPTION:
Long-term benefits of statins on prevention of cardiovascular events have been consistently shown in several populations. It has been demonstrated that, with particular regard to subjects at high risk, the lower LDL-cholesterol levels, the lower the incidence of cardiovascular outcomes. Beneficial effects of statins can be attributed to their lipid-lowering ability as well as to additional benefits. The so-called pleiotropic effects on low grade inflammation status have been described in subsets of subjects with different cardiovascular profiles. The most common inflammatory marker used in clinical practice is the high-sensitivity C-reactive protein (CRP) level, but a number of others has also been investigated.

Disturbances of glucose metabolism accompanied by insulin resistance are pro-inflammatory conditions which may accelerate atherosclerosis. Diabetic populations are at high cardiovascular risk and strict control of lipoprotein concentrations is recommended. Several recent studies showed the efficacy of statins on primary and secondary prevention of cardiovascular events in diabetic populations. The goal of 100 mg/dL for LDL-cholesterol may be too elevated for subjects at very high risk for whom a target of 70 mg/dl has been suggested. High statin doses may be necessary, which increases its adverse effects. Given that statin monotherapy may be insufficient for the desirable reduction in LDL levels, a combination of lipid-lowering agents has become frequent in clinical practice. In particular, statin and ezetimibe combination has been shown to be very effective in reducing total and LDL cholesterol levels.

Ezetimibe is a specific cholesterol absorption inhibitor that acts at the brush border of the small intestine, blocking the absorption of dietary and biliary cholesterol and plant sterols, resulting in intracellular cholesterol depletion via the Niemann-Pick C1-like transporter. Adding ezetimibe to statin therapy induces a 15% reduction in LDL levels compared with only 6% achieved by doubling the dose of statins. Data concerning the pleiotropic effects of this combination are controversial. One study, in which CRP level was used as the inflammatory marker, found that a combination of simvastatin and ezetimibe produced an incremental effect in lowering CRP, independently of the improvement in lipoprotein concentrations. Although few studies have confirmed this finding, as far as we know, data regarding simvastatin-ezetimibe combination induced-changes in serum interleukin-6 (IL-6) and tumor necrosis factor alpha (TNF-a) levels are lacking. We tested the hypothesis that this combination would induce improvement in inflammatory status, as reflected by leukocyte count and CRP, IL-6 and TNF-α levels.

Therefore, this study evaluates whether the combination of lipid-lowering effects of low-to-moderate dose of simvastatin and ezetimibe also results in a synergistic effect that reduces the pro-inflammatory status of pre-diabetic subjects with mild-to-moderate hypercholesterolemia.

Subjects and Methods:

Participants were selected from the Federal University of São Paulo outpatient clinics. The study was approved by the institutional ethical committee and all participants were provided with written informed consent.

Eligible subjects were men and women, aged from 18 to 75 years, with a body mass index (BMI) ranging from 25 to 40 kg/m2 and pre-diabetes (impaired glucose tolerance or impaired fasting glucose). Entry criteria required triglyceride levels ≤ 350 mg/dl and LDL cholesterol ≤ 200 mg/dl, stable blood pressure and no evidence of cardiovascular, hepatic or renal diseases. Subjects were not taking anti-inflammatory agents or others interfering with lipid or glucose metabolism. Eligible participants were recruited from June 2005 to May 2006. Two-hundred-ninety subjects with weight excess, with or without family history of diabetes, were screened for the interventional protocol and 50 with impaired glucose tolerance (IGT) or impaired fasting glucose (IFG) were randomly assigned to 2 groups that would receive ezetimibe 10 mg/d (n = 25) or simvastatin 20 mg/d (n = 25), preceded by a 2-week run-in period. Monotherapies were maintained for 12 weeks; thereafter the drugs were combined in each group for an additional 12-week period. All participants received individual counseling for a healthy lifestyle and had monthly visits. Treatment was to be discontinued prematurely if transaminases exceeded 3 times the upper limit of reference or creatine phosphokinase (CPK) 10 times, but no subject met these criteria. One of the ezetimibe group dropped out due to non-compliance.

Baseline, 12-week and 24-week blood samples were drawn in the morning, after a 12-hour fast, for glucose, lipid profile, including apolipoprotein A-I and B, leukocyte count and inflammatory markers were made. A LDL-cholesterol goal of 100 mg/dl was used in the present study (8,22).

Laboratory analysis: Plasma glucose, transaminases, CPK and creatinine were determined by routine methods. Serum lipid levels (total cholesterol, HDL-cholesterol, and triglycerides) were analyzed by commercially available tests (Roche Diagnostics GmbH, Mannheim, Germany). Blood samples were stored at -20ºC until determinations of apolipoproteins and inflammatory markers. Apolipoprotein A-I and B were measured by immunoturbidimetry (Olympus Life and Material Science Europa GmbH, Lismeeham, Ireland), with an intra-assay coefficient of variability (CV) of 1.26-1.30% and 0.93-1.17% respectively, and an inter-assay CV of 1.43-1.55% and 1.10-1.46%, respectively. High-sensitivity CRP (Immulite - DPC, Los Angeles, CA, USA), TNF-α and IL-6 (Immulite - Euro/DPC, Llanberis, Gwynedd, UK) were determined by chemiluminescent immunometric assay. The sensitivity of CRP assay was 0.01 mg/dL (intra-assay CV 4.2-6.4% and inter-assay CV 4.8-10%), of TNF-α assay 1.7 pg/mL (intra-assay CV 2.6-3.6%, inter-assay CV 4.0-6.5%) and of IL-6 assay was 2.0 pg/mL (intra-assay CV 3.5-6.2%, inter-assay CV 5.1-7.5%).

Statistical analysis: Data were expressed as mean values and standard errors or deviations. Unpaired Student's t test was used to compare groups at baseline and chi-square to assess differences between qualitative data. One-way ANOVA for repeated measures was used to evaluate the effect of drugs over time and to compare data between groups of subjects according to the type of therapy. Pairwise contrasts were made by comparing least-square mean estimates, and P values adjusted for multiple comparisons using the Bonferroni Holm method. The level of significance was set at P < 0.05. Correlation between variables was tested by the Pearson coefficient, also employed to assess whether changes in variables over time were correlated. Data analysis was performed using Statistical Analysis System software, version 8.2 (SAS Institute, Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

* Both sexes, aged from 18 to 75 years, with a body mass index ranging from 25 to 40 kg/m2 and pre-diabetes (impaired glucose tolerance or impaired fasting glucose).

Exclusion Criteria:

* Blood triglyceride concentration >350 mg/dl and LDL cholesterol >200 mg/dl, unstable blood pressure, clinical evidences of cardiovascular, hepatic or renal diseases, use of anti-inflammatory agents or others interfering with lipid or glucose metabolism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-06; Primary Completion 2006-05 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
C reactive protein | Serum C reactive protein was detected at baseline, before starting monotherapy with simvastatin or ezetimibe, and after 12 weeks of each monotherapy
  CRP is one of the most important inflammatory marker and its determination has been considered a non-traditional risk factor for several chronic diseases including diabetes and cardiovascular diseases.
C reactive protein | C reactive protein (CRP) concentration was determined after 12 weeks of monotherapy (simvastatin or ezetimibe) and was compared with the concentration after more 12 weeks of combined therapy
  CRP is one of the most important inflammatory marker and its determination has been considered a non-traditional risk factor for several chronic diseases including diabetes and cardiovascular diseases.
C reactive protein | Serum C reactive protein (CRP) concentration detected at baseline was compared with that obtained after of combined therapy of simvastatin plus ezetimibe (week 24)
  CRP is one of the most important inflammatory marker and its determination has been considered a non-traditional risk factor for several chronic diseases including diabetes and cardiovascular diseases.

SECONDARY OUTCOMES:
Interleukin-6 | Circulating interleukin-6 concentration was determined at baseline (before monotherapy with simvastatin or ezetimibe) and after a 12-week period of each monotherapy
  Interleukin-6 (IL-6) is a cytokine also produced by the adiposo tissue; its measurement in blood has been used as inflammatory marker for research purposes.
Tumor necrosis factor alpha | Tumor necrosis factor alfa concentration was determined at baseline (before monotherapy with simvastatin or ezetimibe) and after a 12-week period of each monotherapy
  Tumor necrosis factor alfa (TNF-alpha) is secreted by adipose tissue and released to blood. Circulating levels of TNF-alpha may be indicative of a proinflammatory status, which is a initiating mechanism of metabolic and cardiovascular abnormalities.
Interleukin-6 | Interleukin-6 concentration was determined after 12 weeks of monotherapy with simvastatin or ezetimibe and compared with the concentrations after more 12 weeks of combined therapy
  Interleukin-6 (IL-6) is a cytokine also produced by the adiposo tissue; its measurement in blood has been used as inflammatory marker for research purposes.
Tumor Necrosis Factor Alpha | Serum tumor necrosis factor alpha concentration was determined after 12 weeks of monotherapy with simvastatin or ezetimibe and compared with the concentrations after more 12 weeks of combined therapy
  Tumor necrosis factor alfa (TNF-alpha) is secreted by adipose tissue and released to blood. Circulating levels of TNF-alpha may be indicative of a proinflammatory status, which is a initiating mechanism of metabolic and cardiovascular abnormalities.
Interleukin-6 | Interleukin-6 concentration detected at baseline was compared with that obtained after of combined therapy of simvastatin plus ezetimibe (week 24)
  nterleukin-6 (IL-6) is a cytokine also produced by the adiposo tissue; its measurement in blood has been used as inflammatory marker for research purposes.
Tumor necrosis factor alpha | Tumor necrosis factor alpha concentration detected at baseline was compared with that obtained after of combined therapy of simvastatin plus ezetimibe (week 24)
  Tumor necrosis factor alfa (TNF-alpha) is secreted by adipose tissue and released to blood. Circulating levels of TNF-alpha may be indicative of a proinflammatory status, which is a initiating mechanism of metabolic and cardiovascular abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra RG Ferreira, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Hospital do Rim e Hipertensao da UNIFESP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Kater AL, Batista MC, Ferreira SR. Synergistic effect of simvastatin and ezetimibe on lipid and pro-inflammatory profiles in pre-diabetic subjects. Diabetol Metab Syndr. 2010 Jun 7;2:34. doi: 10.1186/1758-5996-2-34. PMID 20529243